CLINICAL TRIAL: NCT05438485
Title: JUMP, Journey to Understand Methylmalonic Acidemia and Propionic Acidemia - a Natural History Study
Brief Title: Natural History Study of Patients With Methylmalonic Acidemia and Propionic Acidemia
Acronym: JUMP
Status: Terminated | Type: Observational
Why Stopped: The decision to terminate the study was based on business considerations by the Sponsor.
Sponsor: HemoShear Therapeutics (Industry)
Collaborators: AllStripes Research Inc. (Industry); Prometrika, LLC (Industry); Genome Medical (Unknown)
Responsible Party: Sponsor
Other Study IDs: HST21-NH03
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2022-09

CONDITIONS: Methylmalonic Acidemia; Propionic Acidemia
Keywords: Methylmalonic Acidemia; Propionic Acidemia; Organic Acidemia; Inborn errors of metabolism; PCCA; PCCB; Propionyl-coenzyme A carboxylase; MMUT; Methylmalonyl-CoA mutase; Metabolic disease; Genetic disease; HemoShear; Natural History Study; JUMP
MeSH Terms: conditions — Methylmalonic acidemia; Propionic Acidemia; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methylmalonic Acidemia (MMA): Approximately 60 subjects with Methylmalonic Acidemia
  Interventions: Other: Registry
- Propionic Acidemia (PA): Approximately 60 subjects with Propionic Acidemia
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Observational (Registry)

SUMMARY:
The JUMP (Journey to Understand MMA and PA) Study is being conducted by HemoShear Therapeutics and AllStripes, a rare disease online research platform. JUMP is designed to accelerate understanding of the natural course of methylmalonic acidemia (MMA) and propionic acidemia (PA) disease and treatment for families, researchers, clinicians and industry.

The study will collect and provide patient medical record information from multiple institutions for families to access in one place at no cost. AllStripes will remove identifying information like name and address from these medical records and aggregate this data for the HemoShear team to better understand the medical experience and progression of MMA and PA over time. In addition, academic researchers, healthcare practitioners and patient advocacy groups can apply to use the collective patient community data to answer specific research questions at no cost.

HemoShear is collecting natural history data on MMA and PA because the company needs insight into the real-world experience of many patients to better understand the disease and be able to scientifically demonstrate whether the potential new treatment they are developing is effective in improving outcomes.

This natural history study will include retrospective and prospective components. The retrospective component will consist of data abstracted from primarily electronic health records (eHR) and some paper records. The prospective component will include ongoing collection of medical records from enrolled participants, and participants may opt in to complete health-related questionnaires and an optional genetic testing sub-study.

After signing informed consent, participants or their legal guardians will grant permission to AllStripes to collect their health records for data abstraction.

Participants may opt into an optional no cost genetic testing sub-study. The JUMP (Journey to Understand MMA and PA) sub-study will help assess whether the genetic variant of the affected person may relate to disease severity and treatment response. Getting genetic testing will enable participants to understand the genetic mutation that causes their type of methylmalonic acidemia (MMA) or propionic acidemia (PA). Knowing the genetic mutations (whether from the MMUT, MMAA or MMAB gene or PCCA or PCCB) can help the impacted person, their caregivers and healthcare professionals understand the potential course of disease and select approaches to better manage the disease. The additional information will enable HemoShear and AllStripes to understand whether different genetic variants impact the disease journey and outcomes.

A separate informed consent will be obtained for participating in the sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or participant's legal guardian must provide signed, informed eConsent/eAssent prior to releasing health records or performing any study-related procedures.
2. Confirmed diagnosis of MMA or PA.
3. Reside in the US, Canada, or United Kingdom and have all medical records available for abstraction.

Exclusion Criteria:

1. Participant or participant's legal guardian is unable to provide complete access to medical records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 120 participants will be enrolled from the United States, Canada, and the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Understanding of the natural course of methylmalonic acidemia (MMA) and propionic acidemia (PA) disease and treatment for families, researchers, clinicians and industry. | 5 years

CONTACTS AND LOCATIONS:
Locations (3):
- AllStripes, San Francisco, California, United States
- AllStripes, Remote, Remote, Canada
- AllStripes, Remote, Remote, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to information about participation in JUMP — https://www.allstripes.com/study/jump
- See also: Link to information about optional genetic testing. Only participants in JUMP will receive link to optional genetic testing. — https://www.genomemedical.com/programs/hemoshear/
- See also: Link to information about participation in JUMP for MMA — https://www.allstripes.com/mma
- See also: Link to information about participation in JUMP for PA — https://www.allstripes.com/pa